CLINICAL TRIAL: NCT02707978
Title: F 18 T807 Tau PET Imaging of Frontotemporal Dementia
Brief Title: F 18 T807 Tau PET Imaging of Frontotemporal Dementia (FTD)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Problems with contracts .
Sponsor: Tammie L. S. Benzinger, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Tammie L. S. Benzinger, MD, PhD, Associate Professor of Radiology and Neurological Surgery, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IND 123119 Protocol C
Record Dates: First submitted 2015-04-07; First posted 2016-03-14 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease
Keywords: Dementia; Brain Diseases; Central Nervous System Diseases; Mild Cognitive Impairment; tauopathies; Neurodegenerative Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Cognitive Dysfunction; Tauopathies; Neurodegenerative Diseases | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental F 18 T807 (Experimental)
  Interventions: Drug: F 18 T807

INTERVENTIONS:
Drug: F 18 T807 — Participants will receive a single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807. For those who cannot tolerate the full exam, participants will receive single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807.
  Other Names: 18F-AV-1451

SUMMARY:
The purpose of this research study is to evaluate tau distribution in the brain of subjects with: FTD caused by different genetic mutations, any mutation carriers (with or without symptoms), any non-mutation carrier, any sporadic FTD, normal controls.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, at least 18 years of age.
2. Clinically diagnosed with frontotemporal dementia (FTD), or a carrier of a mutation known to cause FTD (with or without symptoms); or a normal control.
3. Participant is able and willing to undergo testing (MRI or CT, PET, radioactive tracer injection, LP; for those unable to undergo an MRI, CT will be used to generate regions-of-interest).
4. Pre-menopausal women will have a negative a urine pregnancy test within 24 hours of T807 drug administration.

Exclusion Criteria:

1. Has any condition that, in the Investigator's opinion, could increase risk to the participant, limit the participant's ability to tolerate the experimental procedures, or interfere with the collection/analysis of the data (for example, participants with severe chronic back pain might not be able to lie still during the scanning procedures).
2. Is deemed likely unable to perform the imaging procedures for any reason.
3. Has a history of Torsades de Pointes or is taking medications known to prolong QT interval. To determine who will be excluded from this study based on this criterion, we will review participant's medical history and current medications at time of screening. Participants will be excluded from the study if any of the following restricted medications are being taken:

   * Disopyramide
   * Dofetilide
   * Ibutilide
   * Procainamide
   * Quinidine
   * Sotalol
   * Bepridil
4. Has hypersensitivity to F 18 T807 or any of its excipients.
5. Contraindications to PET, PET-CT or MR (e.g. electronic medical devices, inability to lie still for long periods) that make it unsafe for the individual to participate.
6. Severe claustrophobia.
7. Currently pregnant or breast-feeding.
8. For those electing to undergo the optional lumbar puncture: on

anticoagulant of any form prior to lumbar puncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-30 (Estimated); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
F 18 T807 Standard Uptake Value Ratios (SUVR) will be correlated with other imaging modalities (MRI, PET amyloid imaging) and cognitive performance. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States